CLINICAL TRIAL: NCT03853148
Title: Activate For Life: A Nurse Delivered Hybrid Telehealth/mHealth Aging In Place Intervention To Address Pain And Fatigue In Low-income Older Adults
Brief Title: Activate For Life: mHealth Intervention To Address Pain And Fatigue In Low-income Older Adults Aging In Place
Acronym: Activate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Teresa Kelechi, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pr00076835; 5P20NR016575-05 (NIH)
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Results first posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Pain, Chronic; Fatigue Syndrome, Chronic; Aging
MeSH Terms: conditions — Chronic Pain; Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Otago (Active Comparator): The Otago exercise program consists of the following: 1) A series of warm-up exercises, 2) Select exercises from the 17 Otago exercises which challenge the participant's strength and balance for up to 30 minutes, three times a week, 3) A walking program for up to 30 minutes, three times a week. Each Otago will be tailored for each participant's ability level.
  Interventions: Behavioral: Otago
- Otago + Gentle yogic breathing (Active Comparator): The GYYB is a one-hour program containing gentle physical Yoga postures that participants could practice sitting on a chair for 30 minutes. These exercises are designed based on improving the overall flexibility, bodily control and mindfulness in movements. Following the gentle yoga postures, the participants will perform Yogic breathing exercises for 30 minutes. These exercises are known to promote relaxation, mood, pain and anxiety scores that are highly relevant to the target population and are reported to stimulate measurable biomarker changes in the saliva. During the in-person session the Yoga instructor will explain the GYYB program to participants in the Otago+GYYB group each exercise and their perceived benefits.
  Interventions: Behavioral: Otago; Behavioral: Gentle yogic breathing
- Otago + GYYB + Behavioral activation (Active Comparator): This condition will incorporate Otago and GYYB as above and will also include behavioral activation to address motivation and affect. Behavioral Activation incorporates daily planners and worksheets to identify and rate reinforcing behaviors and is often used in conjunction with other interventions because components of these interventions are easily incorporated into the daily planner based activities. Each participant outlines general values and specific behaviors that 'demonstrate' each value, compiling a list of the latter. This list is then used to generate 10 to 20 highly defined values-based, reinforcing activities. Next, this list is combined with the activities outlines in Otago and GYYB and this master list is used to schedule these values-based activities for the next two days.
  Interventions: Behavioral: Otago; Behavioral: Gentle yogic breathing; Behavioral: Behavioral Activation
- Caregiver Gentle yoga & yogic breathing (Experimental): The GYYB is a one-hour program containing gentle physical Yoga postures that participants could practice sitting on a chair for 30 minutes. These exercises are designed based on improving the overall flexibility, bodily control and mindfulness in movements. Following the gentle yoga postures, the participants will perform Yogic breathing exercises for 30 minutes. These exercises are known to promote relaxation, mood, pain and anxiety scores that are highly relevant to the target population and are reported to stimulate measurable biomarker changes in the saliva. During the in-person session the Yoga instructor will explain the GYYB program to participants in the GYYB group each exercise and their perceived benefits.
  Interventions: Behavioral: Caregiver Gentle yogic breathing

INTERVENTIONS:
Behavioral: Otago — Exercise program for strength and balance
  Arms: Otago; Otago + GYYB + Behavioral activation; Otago + Gentle yogic breathing
Behavioral: Gentle yogic breathing — yogic breathing
  Other Names: GYYB
  Arms: Otago + GYYB + Behavioral activation; Otago + Gentle yogic breathing
Behavioral: Behavioral Activation — Behavioral Activation incorporates daily planners and worksheets to identify and rate reinforcing behaviors and is often used in conjunction with other interventions because components of these interventions are easily incorporated into the daily planner based activities.
  Arms: Otago + GYYB + Behavioral activation
Behavioral: Caregiver Gentle yogic breathing — yogic breathing
  Other Names: Caregiver GYYB
  Arms: Caregiver Gentle yoga & yogic breathing

SUMMARY:
The Overall Aim of the present proposal is to evaluate the feasibility of an integrated mind-body intervention, Activate for Life, to improve overall physical activity and mental health and reduce pain and fatigue, resulting in increased likelihood of Aging in Place. Both subjective self-report (i.e., Patient-Reported Outcomes Measurement Information System PROMIS measures of pain, fatigue, depression and anxiety) and objective accelerometer data will be collected, along with standardized measures of balance, strength, and stability. In addition, the measures will be complemented with biomarker-based measures of stress, including cortisol based and 1,5-AG anhydroglucitol assays before, during, and after treatment that are correlated with stress, and fatigue symptoms.

DETAILED DESCRIPTION:
The goal of supplement study is to test the feasibility of a self-managed (SM), electronic/mobile Health (e/mHealth) yoga intervention for reducing stress symptoms (burden) in older caregivers (CG) of people with Alzheimer's Disease and related dementia's (PWD). CG burden can exacerbate a myriad of physical and psychosocial comorbidities in CGs as well as PWD neuropsychiatric symptoms. These effects may be further amplified in older CG with underlying health concerns or those who are not able to access programs for effective management of their own medical or self-care needs. Low-impact physical activities such as gentle Yoga (GY) have shown positive effects on mood and symptoms of pain and fatigue in older community dwellers, and digital e/mHealth platforms have a great deal of potential to overcome financial and medical barriers for the delivery SM stress interventions across demographic boundaries. In this study, we will examine the feasibility of a 12-week e/mHealth gentle yoga+yogic breathing (GYYB) intervention for alleviating symptoms of burden in aging CG of PWD (Aim 1); measure initial changes in stress and QoL indicators in CG and PWD (post- vs. pre-intervention) to inform an adequately-powered, future efficacy trial (Aim 2), and; establish a Dyadic Analysis Training Program for Medical University of South Carolina (MUSC) faculty within the College of Nursing and P20 Symptom Self-Management Center (SSMC) to support future research evaluating the influence of care-recipient interactions on health outcomes (Aim 3). Feasibility will be assessed using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework, and will include measures such as recruitment, adherence, treatment satisfaction, attrition, and feedback for intervention refinement. Data related to CG physical function, fatigue, depression, social isolation, loneliness, relationship quality, burden, and stress biomarkers, as well as PWD and CG QoL, will be collected via daily electronic practice logs and interviews at study beginning and end. Older (45 yrs. old and older) male and female CG (N=20) of PWD regularly attending respite care (RCC) programs will be recruited from an existing study population (R01 NR016466) participating in CG-RCC mealtime partnerships for improved PWD nutritional outcomes. The HIPAA-compliant GYYB intervention will employ 'tablets' that allow CG to practice GYYB at home by following along with recorded lessons. CG will initially be trained on the use of the tablet and proper GYYB practices by the study coordinator (in-home), with weekly follow up (videoconference/phone) for the duration of the study. This investigation is ideally aligned with the aims of the parent SSMC (P20 NR016575) that are focused on providing infrastructure and community-based resources for design and ecologically-valid testing of self management (SM) interventions for individuals with chronic conditions.

ELIGIBILITY:
Inclusion and Exclusion Criteria for Older Adults (Arms 1, 2, 3):

* Males and females older adults 60 years of age and older living in a Humanities Foundation apartment complex or in their own homes
* PROMIS pain interference score of eight or above and/or a PROMIS pain behavior score of 15 or above (for older adults)
* Able to ambulate 150 feet with or without the use of an assistive device
* Able to follow simple instructions
* Able to read, speak, and write English,
* Able to operate tablet device and wearable activity tracker,
* Not currently enrolled in an exercise program.

Exclusion Criteria:

* Inability or unwillingness of participant to give informed consent,
* Physical, cognitive, sensory or psychiatric disability that would limit participants from engaging in self-management program as noted by a Mini-Cog score of 0-2.
* Unwillingness to wear a physical activity tracker during the course of the study.

Inclusion and Exclusion Criteria for Caregivers (Arm 4)

* CG must be able to speak and read English
* CG must be 45 years of age or older
* CG must be able to provide consent for himself or herself
* CG must live with or on same property as the PWD
* CG be primarily responsible for care provision of the PWD in the home (i.e., is not paid for services; provides 4 hours or more of care/day; assists with activities of daily living-ADLs)

Exclusion Criteria:

* CG for whom yoga techniques would be detrimental due to physical limitations,
* CG who are enrolled in other Yoga-related clinical trials, or who are currently engaged in regular Yoga activity once per week or more.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- College of Nursing Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kelechi TJ, Layne D, Mueller M, Madisetti M, Balasubramanian S. Feasibility and Preliminary Impact of a Web-Based Mind Body Intervention for Older Dementia Caregivers. West J Nurs Res. 2024 Jun;46(6):416-427. doi: 10.1177/01939459241247926. Epub 2024 Apr 24. PMID 38655852
- [Derived] Hernandez-Tejada MA, Nagel A, Madisetti M, Balasubramanian S, Kelechi T. Feasibility trial of an integrated treatment "Activate for Life" for physical and mental well-being in older adults. Pilot Feasibility Stud. 2022 Feb 11;8(1):38. doi: 10.1186/s40814-022-01000-8. PMID 35148798

RESULTS

PARTICIPANT FLOW:
Groups:
- Otago + GYYB + Behavioral Activation: This condition will incorporate OEP and GYYB as above and will also include behavioral activation to address motivation and affect. Behavioral Activation incorporates daily planners and worksheets to identify and rate reinforcing behaviors and is often used in conjunction with other interventions because components of these interventions are easily incorporated into the daily planner based activities. Each participant outlines general values and specific behaviors that 'demonstrate' each value, compiling a list of the latter. This list is then used to generate 10 to 20 highly defined values-based, reinforcing activities. Next, this list is combined with the activities outlines in Otago and GYYB and this master list is used to schedule these values-based activities for the next two days.
  Otago: Exercise program for strength and balance
  Gentle yogic breathing: yogic breathing
  Behavioral Activation: Behavioral Activation incorporates daily planners and worksheets to identify and rate reinforcing behaviors and is often used in conjunction with other interventions because components of these interventions are easily incorporated into the daily planner based activities.
Period: Overall Study
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Started | 10 | 10 | 10 | 20
Completed (The participant "completers" varied throughout the study for each of the outcomes which ranged from 8 completers to as low as 2 completers, depending on the outcome. Reported in the Not Completed section here are the lowest numbers of completers in any one outcome.) | 5 | 2 | 2 | 15
Not Completed | 5 | 8 | 8 | 5
Not completed — Did not fill in or incomplete questionnaire; missing data; could not score questionnaire, | 5 | 8 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing | Total
Number analyzed (Participants) | 10 | 10 | 10 | 20 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 2 | 8 | 13
  >=65 years | 10 | 7 | 8 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.4 (5.6) | 68.5 (7.5) | 69.8 (5.4) | 68.7 (8.0) | 70.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 7 | 14 | 35
  Male | 3 | 3 | 3 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 20 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 8 | 2 | 20
  White | 5 | 5 | 2 | 18 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 20 | 50

OUTCOME MEASURES:

1. Primary Outcome: Older Adult Pain Intensity
Description: Change in mean pain T-scores as measured with the Patient-Reported Outcomes Measurement Information System PROMIS Pain Intensity short form 3a, which allows for individuals to report how much a person hurts. The lowest possible raw score is 4; the highest possible raw score is 20. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the higher above 50 the more pain interferes with aspects of one's life compared to the general population. Scores <55 within normal limits, 55-60 mild, 61-70 moderate, >70 severe pain intensity.
Time Frame: Baseline to 12 weeks
Population: This questionnaire was given to the older adults only, not the caregivers.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 8 | 6 | 4 | 0
T-score | -3.25 (0.3) | -2.8 (4.2) | -0.5 (1.6) |

2. Primary Outcome: Older Adult Fatigue
Description: Change in mean fatigue T-score as measured by PROMIS Fatigue short form 6a, 6 items that assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. The lowest possible raw score is 6; the highest possible raw score is 30. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the higher above 50 the worse the fatigue the individual has compared to the general population. Scores <55 within normal limits, 55-60 mild, 61-70 moderate, >70 severe fatigue.
Time Frame: Baseline to 12 weeks
Population: This questionnaire was given to the older adults only, not the caregivers.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 8 | 5 | 5 | 0
T-score | 0.9 (1.5) | -0.8 (7.6) | -4.0 (1.9) |

3. Primary Outcome: Older Adult Pain Behavior
Description: Change in mean pain T-score as measured with PROMIS Pain Behavior short form 7a, which allows for self-reported external manifestations of pain: behaviors that typically indicate to others that an individual is experiencing pain. These actions or reactions can be verbal or nonverbal, and involuntary or deliberate. The lowest possible raw score is 7; the highest possible raw score is 42. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the higher above 50 the worse or more pain behavior the individual has compared to the general population. Scores <55 within normal limits, 55-60 mild, 61-70 moderate, >70 severe pain behavior.
Time Frame: Baseline to 12 weeks
Population: This questionnaire was given to the older adults only, not the caregivers.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 7 | 6 | 4 | 0
T-score | -0.7 (1.2) | 2.2 (6.1) | -3.7 (1.7) |

4. Secondary Outcome: Older Adult Functional Status
Description: Change in mean functional T-score as measured by PROMIS Physical Function 10b, 10-item instrument that assesses sit-to-stand, walking, and balance abilities as well as self-reported physical abilities including mobility, upper and lower extremity strength, core strength, and activities of daily living. The lowest possible raw score is 10; the highest possible raw score is 50. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the lower scores below 10 indicate a greater degree of impaired function. Scores >55 within normal limits, 56-40 mild, 41-30 moderate, <30 severe (worse functional status).
Time Frame: Baseline to 12 weeks
Population: This questionnaire was completed by both older adults and caregivers.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 7 | 5 | 4 | 15
T-score | 1.0 (4) | 3.1 (1.5) | 1.5 (2.1) | 1.7 (0.8)

5. Secondary Outcome: Older Adult Balance
Description: Change in mean balance scores measured with the Berg Balance Scale, which includes 14 tests (e.g., standing on one leg, stepping over obstacles). Each task is worth 0-2 points and points are summed for a total score. Higher scores indicate better balance and lower scores indicate fall risk. Scores range from 0 - 56. 1 - 20 indicates a person will likely need assistance of a wheelchair to move around safety due to major limitations/poor balance noted during the assessment of the tasks; 21 - 40 indicates a person will need some type of walking assistance such as a cane or walker due to problems or limitations with some of the movement on the scale; 41 - 56 indicates a person is considered independent and able to move around safely without assistance and is at low risk for falling.
Time Frame: Baseline to 12 weeks
Population: This questionnaire was given to the older adults only, not the caregivers.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 6 | 2 | 2 | 0
Score on a scale | -1.8 (1.1) | -4.5 (0.7) | -4.5 (0.3) |

6. Secondary Outcome: Older Adult Sit-to-Stand Capability
Description: Change in mean number of times an individual comes to a full standing position from the seated position when 30 seconds have elapsed measured with the 30-Second (s) Chair Test to assess lower body strength. Higher numbers indicate better lower body strength. Below average sit-to-stand scores per age groups are as follows: men 60-64 <14, women < 12; men 65-69 <12, women <11; men 70-74 <12; women <10; men 75-79 <11, women <10; men 81-84 <10, women <9; men 85-89 <8, women <8; men 90-94 <7, women <4. Unfortunately we were unable to collect these data due to COVID restrictions. We were unable to make home visits or have participants come into our research clinic to assess their sit-to-stand ability because we were not permitted to have patient contact.
Time Frame: Baseline to 12 weeks
Population: We were unable to collect these data due to coronavirus disease of 2019 (COVID-19) restrictions. We were unable to make home visits or have participants come into our research clinic to assess their sit-to-stand ability because we were not permitted to have patient contact.
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Older Adult Walking Ability
Description: Change in mean walking distance in feet over a timed two-minute period measured with the Two-Minute Walk Test to assess walking ability.
Time Frame: Baseline to 12 weeks
Population: This questionnaire was given to the older adults only, not the caregivers.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 7 | 5 | 4 | 0
Feet | 17.4 (17.1) | -6.8 (3) | 24 (15.8) |

8. Secondary Outcome: Older Adult Depression
Description: Change in mean depression T-score measured with the Patient-Reported Outcomes Measurement Information System PROMIS Depression short form 8a, 8 individual items allow for different responses which are scored separately to provide specific information about self-reported negative mood (sadness, guilt), view of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation) as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). The lowest possible raw score is 8; the highest possible raw score is 40. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the higher above 50 suggests an individual has greater depressive symptoms compared to the general population.
Time Frame: Baseline to 12 weeks
Population: This questionnaire was given to the older adults only, not the caregivers.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 8 | 6 | 5 | 0
T-score | -1.57 (0.52) | 0.37 (0.36) | -5.26 (2.06) |

9. Secondary Outcome: Older Adult Self Efficacy
Description: Change in mean self efficacy score measured with the Common Data Repository For Nursing Science (cdRNS) National Institute of Nursing Research, Self-Efficacy for Managing Chronic Disease questionnaire which contains 6-items that cover several domains that are common across many chronic diseases including symptom control, role function, emotional functioning and communicating with physicians. Scores range from 1 (not at all confident) to 10 (totally confident). A sum score is reported. Higher score indicate higher self efficacy or confidence in managing one's disease.
Time Frame: Baseline to 12 weeks
Population: This questionnaire was given to the older adults only, not the caregivers.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 8 | 6 | 5 | 0
Score on a scale | -0.39 (0.95) | 0.06 (0.59) | -0.31 (0.32) |

10. Secondary Outcome: Older Adult Daily Steps
Description: Steps were measured with an actigraph and reported as mean numbers of steps taken per week during the 12-week study period. The mean number of steps per week for the participants who completed the study in each arm is reported for the 12-week final study measurement period. Full range of steps taken is reported indicating minimum and maximum steps taken at the end of study 12-week period for the participants who completed all 12 weeks of the study.
Time Frame: Baseline to 12 weeks
Population: Steps taken were only measured in older adults only, not the caregivers.
Measure: Mean (Full Range); unit: Steps walked
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 5 | 3 | 4 | 0
Steps walked | 32201 [5130 to 90057] | 29577 [15693 to 46431] | 24699 [15499 to 35805] |

11. Secondary Outcome: Caregiver Anxiety
Description: Change in mean anxiety status T-score measured with PROMIS Anxiety short form 6a, 6 individual items allow for different responses which are scored separately to provide specific information about self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). The lowest possible raw score is 6; the highest possible raw score is 30. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the higher above 50 suggests an individual has greater anxiety symptoms compared to the general population. Scores <55 within normal limits, 55-60 mild, 61-70 moderate, >70 severe anxiety.
Time Frame: Baseline to 12 weeks
Population: Anxiety was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
T-score |  |  |  | 1.7 [-3.8 to 7.3]

12. Secondary Outcome: Caregiver Health Status
Description: Change in mean health status score measured with PROMIS Global Health Scale, 10 individual items allow for different responses which are scored separately to provide specific information about perceptions of physical function, pain, fatigue, emotional distress, social health and general perceptions of health. The lowest possible raw score is 4; the highest possible raw score is 20. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the higher above 50 the better or more healthy the individual is compared to the general population. Scores 20-35 = poor, 36-42 fair, 43-50 good, 51-57 very good, >58 excellent health status.
Time Frame: Baseline to 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
T-score |  |  |  | 1.2 [-0.4 to 2.8]

13. Secondary Outcome: Caregiver Functional Health
Description: Change in mean functional health T-score measured with PROMIS Physical Function Scale short form 8b, 8 individual items allow for different responses which are scored separately to provide specific information about self-reported current capability rather than actual performance of physical activities. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the higher above 50 the better function the individual has compared to the general population. Scores >55 within normal limits, 56-40 mild, 41-30 moderate, <30 severe physical functional impairment (worse health).
Time Frame: Baseline to 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
T-score |  |  |  | 1.7 [-1.7 to 5.0]

14. Secondary Outcome: Caregiver Sleep Disturbance
Description: Change in mean sleep disturbance score measured with PROMIS Sleep Disturbance short form 6a, 6 individual items allow for different responses which are scored separately to provide specific information about self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. The lowest possible raw score is 6; the highest possible raw score is 30. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the higher above 50 the worse or the greater the individual's sleep is disturbed compared to individuals with chronic conditions. Scores <55 within normal limits, 55-60 mild, 61-70 moderate, >70 severe sleep disturbance.
Time Frame: Baseline to 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
T-score |  |  |  | -0.6 [-3.8 to 2.7]

15. Secondary Outcome: Caregiver Depression
Description: Change in mean depression score measured with PROMIS Depression short form 8a, 8 individual items allow for different responses which are scored separately to provide specific information about self-reported negative mood (sadness, guilt), view of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation) as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). The lowest possible raw score is 8; the highest possible raw score is 40. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the higher above 50 suggests an individual has greater depressive symptoms compared to the general population. Scores <55 within normal limits, 55-60 mild, 61-70 moderate, >70 severe depression.
Time Frame: Baseline to 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
T-score |  |  |  | -0.8 [-3.7 to 2.1]

16. Secondary Outcome: Caregiver Depression CES-D
Description: Change in mean depression score measured with the Center for Epidemiological Studies-Depression scale (CES-D), 20 items - that asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms. The cutoff scores (e.g., 16 or greater) identify individuals at risk for clinical depression.
Time Frame: Baseline to 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
Score on a scale |  |  |  | -0.3 [-2.6 to 2.0]

17. Secondary Outcome: Caregiver Fatigue
Description: Change in mean fatigue score measured with the PROMIS Fatigue short form 6a, 6 items that assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. The lowest possible raw score is 6; the highest possible raw score is 30. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the higher above 50 the worse the fatigue the individual has compared to the general population. Scores <55 within normal limits, 55-60 mild, 61-70 moderate, >70 severe fatigue].
Time Frame: Baseline to 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
T-score |  |  |  | -4.7 [-8.2 to -1.1]

18. Secondary Outcome: Caregiver Loneliness
Description: Change in mean loneliness score measured with the University of California Los Angeles UCLA Loneliness Scale which contains 20 items designed to measure one's subjective feelings of loneliness and social isolation. Participants rate each item as either O ("I often feel this way"), S ("I sometimes feel this way"), R ("I rarely feel this way"), N ("I never feel this way"): O's = 3, all S's = 2, all R's = 1, and all N's = 0. Higher scores indicate higher loneliness. Cut-off score of 20 or > indicates loneliness.
Time Frame: Baseline to 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
Score on a scale |  |  |  | -0.9 [-7.2 to 5.3]

19. Secondary Outcome: Caregiver Social Support
Description: Change in mean social support scores measured with the Medical Outcomes Study Social Support Survey Instrument (MOS-SS) contains 19 items with four separate social support subscales and an overall functional social support index. To obtain a score for each subscale, calculate the average of the scores for each item in the subscale. To obtain an overall support index, the average of (1) the scores for all 18 items included in the four subscales, and (2) the score for the one additional item (see last item in the survey) is calculated. Scale scores are transformed to a 0-100 scale and compared to published means reported in Sherbourne, C.D., and Stewart, A.L., "The MOS Social Support Survey,"Social Science and Medicine, 32(6):705-714, 1991. A higher score for an individual scale or for the overall support index indicates more support. Scores suggest poor,(less than 60) fair (60-79) and good social support (more than 80).
Time Frame: 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
Score on a scale |  |  |  | 1.4 [-8.9 to 11.7]

20. Secondary Outcome: Caregiver Burden
Description: Change in mean caregiver burden measured with Zarit Burden Scale (ZBI-12) - 12 items provide a summation score: (0 to 4 points per item, total score range 0 to 48). 0 - 10: no to mild burden; 11 - 20: mild to moderate burden; > 20 high burden.
Time Frame: Baseline to 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
Score on a scale |  |  |  | 3.4 [0.7 to 6.1]

21. Secondary Outcome: Caregiver Quality of Life (QOL)
Description: Change in mean quality of life (QOL) scores measured with the European Quality of Life Five Dimensions (EQ-5D) compromises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and how good/bad one's health with visual analog scale (VAS)) from 0 worst to 100 best health you can imagine) and divided into 3 levels of perceived problems. An EQ-5D summary index is derived by applying a formula that attaches values/weights to each level per dimension. The index is calculated by deducting the appropriate weights from 1, the value for full health and presented as an averaged score. Higher values (scores of 3) indicate extreme pain, depression/anxiety, inability to perform usual activities, unable to wash or dress self, or confined to bed. High VAS scores indicate good perceived health. There are no established/published cut-off scores/values to determine excellent, good, fair or poor QOL levels. Population means are ~70, higher values indicate higher QOL.
Time Frame: Baseline to 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
Score on a scale |  |  |  | -6.3 [-14.7 to 2.2]

22. Secondary Outcome: Caregiver Relationship Quality
Description: Change in mean relationship quality score measured with the Mutuality Scale, a 15-item instrument that measures mutuality (love, shared pleasurable activities, shared values, and reciprocity) from the caregiver perspective. Examples of items are: "How close do you feel to the person you care for?" or "How much do you confide in the person you care for?". Each item is scored on a 5-point Likert-type scale from 0 (not at all), 1 (a little), 2 (some), 3 (quite a bit) to 4 (a great deal). The total scale score, a mean of all item scores, ranges from 0 to 4 (total 0 - 60): higher scores means greater mutuality. There are no established cut-off scores or ranges and are reported in means: 0 = not at all, 1 = a little, 2 = some, 3 = quite a bit, 4 = a great deal.
Time Frame: Baseline to 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
Score on a scale |  |  |  | 0.2 [-0.2 to 0.5]

23. Secondary Outcome: Person With Dementia Quality of Life
Description: Change in mean quality of life score measured with the Life-Alzheimer's Disease (QOL-AD), a 13-item questionnaire designed to be administered via interview to persons with dementia (if able to answer) or by a caregiver. Points are assigned to each item as follows: poor = 1, fair = 2, good = 3, excellent = 4. The total score is the sum of all 13 items. Higher scores indicated higher quality of life. Maximum score is 52. There is no cut-off scores or values/ranges for excellent, good, fair or poor QOL.
Time Frame: Baseline to 12 weeks
Population: Persons with Alzheimer's Disease and Related Dementias, not caregivers or older adults.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
Score on a scale |  |  |  | 1.9 [-2.1 to 5.8]

24. Secondary Outcome: Person With Dementia Activities of Daily Living
Description: Change in mean score on functional activities of daily living measured with the Activities of Daily Living (ADL) Questionnaire which is completed by the caregiver and consists of 46 items for 3 domains: initiation, planning and organization, and performance. The total score, has a range of 0 to 100. The denominator represents the score that would have been obtained if the most severe level of impairment had been indicated for all items rated (excluding those rated ''9''). The numerator represents the total of the actual ratings for all items rated (excluding those rated ''9''). The resultant score represents the level of severity of impairment in ADL. The amount of functional impairment is then rated as ''none to mild'' (0-33),''moderate'' (34-66%), or ''severe'' (.66%). Functional impairment scores are calculated for each subscale individually and for the total of all items. We reported the difference in the total score from baseline to 12-week end of study.
Time Frame: Baseline to 12 weeks
Population: Persons with Alzheimer's Disease and Related Dementias
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
Score on a scale |  |  |  | 1.0 [-2.0 to 4.0]

25. Secondary Outcome: Caregiver of Persons With Dementia Physical Activity
Description: Change in mean minutes (mean difference between baseline and 12 weeks end of study) during the last 7 days engaged in physical activity measured with the International Physical Activity Questionnaire for the Elderly (IPAQ-Short Form) which is comprised of 4 items (sitting, walking, moderate physical activity, vigorous physical activity). For full range (-) indicates fewer mean minutes taken between baseline and 12 weeks.
Time Frame: Baseline to 12 weeks
Population: This was measured in Caregivers of Persons with Alzheimer's Disease and Related Dementias, not older adults.
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 0 | 0 | 0 | 15
Minutes |  |  |  | 213 [-610.5 to 5784.8]

26. Secondary Outcome: Salivary Cortisol
Description: Change in mean laboratory value of cortisol which is an indicator of the hypothalamus-pituitary-adrenal (HPA) axis activity which represents the dominance of the sympathetic nervous system, a measure of psychosomatic stress level. Cortisol reference values are: 3.7-9.5 ng/mL (morning), 1.2-3.0 ng/mL (noon), 0.6-1.9 ng/mL (evening), 0.4-1.0 ng/mL (bedtime). Higher values have been associated with higher stress.
Time Frame: Baseline to 12 weeks
Population: This was measured in both older adults and caregivers of persons with Alzheimer's Disease and Related Dementias.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 7 | 6 | 4 | 15
ng/mL | -0.03 (0.1) | 0.6 (1.4) | -0.5 (1.2) | 2.3 (3.6)

27. Secondary Outcome: Salivary 1,5-Anhydroglucitol (AG)
Description: Change in mean laboratory values of 1,5-Anhydroglucitol (AG) which is a biomarker for glycemic metabolism and is reduced under stressful circumstances. The normal reference value for 1,5 AG is ≥ 14.0 μg/ml.
Time Frame: Baseline to 12 weeks
Population: This was measured in both older adults and caregivers of persons with Alzheimer's Disease and Related Dementias.
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 7 | 6 | 4 | 15
μg/ml | 5.3 (4.8) | 5.4 (5.2) | 3.9 (3.8) | 4.8 (0.6)

28. Secondary Outcome: Adherence
Description: Using study data logs, appropriate use of the interventions was measured by the number of participants who adhered to the protocol for engaging in Arm 1 Otago, Arm 2 Otago + Gentle yoga/yogic breathing, Arm 3 behavioral activation (Older adults) or Arm 4 Gentle yoga/yogic breathing (Caregivers). Adherence was defined as the number of participants (rounded up) who completed the study and were at least 80% adherent to the study protocol for frequency of engaging in the assigned Arm during the 12-week study period.
Time Frame: End of study at 12 weeks post intervention
Population: This was measured in both older adults and caregivers of persons with Alzheimer's Disease and Related Dementias.
Measure: Number; unit: Participants
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
Number analyzed (Participants) | 7 | 6 | 4 | 15
Participants | 6 | 4 | 3 | 7

ADVERSE EVENTS:
Time Frame: From baseline to 12 weeks end of study.
Description: Same definitions used
Arm/Group | Otago | Otago + Gentle Yogic Breathing | Otago + GYYB + Behavioral Activation | Caregiver Gentle Yoga & Yogic Breathing
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 1/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10 | 1/10 | 0/20
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Otago (N=10) | Otago + Gentle Yogic Breathing (N=10) | Otago + GYYB + Behavioral Activation (N=10) | Caregiver Gentle Yoga & Yogic Breathing (N=20)
Fluid buildup around heart (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — One participant self reported through study visit interview
Hospitalization (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant hospitalized due to toxin build up in arm
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant hospitalized for pneumonia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT03853148/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT03853148/SAP_001.pdf
  • Informed Consent Form (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT03853148/ICF_002.pdf